CLINICAL TRIAL: NCT06973785
Title: Non-Narcotic Pain Control After ACL Reconstruction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kurt Spindler, MD, Lead Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-1207
Record Dates: First submitted 2025-03-07; First posted 2025-05-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; ACL Injuries
Keywords: acl; Narcotic use
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Oxycodone; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone- Narcotic (Active Comparator): Arm 1
  Interventions: Drug: Ketorolac
- Ketorolac (Placebo Comparator): Arm 2
  Interventions: Drug: dispense of study drug

INTERVENTIONS:
Drug: dispense of study drug — • Cohort Group 1 (Experimental): ketorolac 10mg with rescue medication oxycodone 5mg All patients will be given acetaminophen
  Other Names: oxycontin
  Arms: Ketorolac
Drug: Ketorolac — Patients will be randomized to either Ketorolac or Oxycodone
  Other Names: Toradol
  Arms: Oxycodone- Narcotic

SUMMARY:
This is a double-blind randomized controlled trial of standard of care therapy, either oral ketorolac (experimental group) or oral oxycodone (control group) to demonstrate efficacy in reducing the percentage of narcotic doses taken and documenting the number of patients with no exposure to any narcotics (take zero oxycodone) after undergoing primary knee ACL reconstruction outpatient surgery.

DETAILED DESCRIPTION:
This is a multi-center, 2 arm, randomized 1:1 controlled trial, with a blinded patient and outcome assessment study. Narcotics are currently the standard of care as part multimodal pain control in major joint surgery including ACLR. Twelve (12) ketorolac (10mg) and twelve (12) oxycodone (5mg) tablets will be shrouded in identical capsules designed for blinding. The capsules will be dispensed in sealed single-pill release blister packets. The enrolled patients will be randomized by the surgeon. The surgeon, clinical team, and patient will be blinded as to treatment (double-blind study). The rescue medication will be specific to each treatment group, encapsulated for blinding, and in a packet labeled RESCUE medication. For the experimental group (ketorolac) they will have 12 oxycodone as rescue medication. For the control group (oxycodone) they will have 12 diclofenac as rescue medication. Both groups will also be given acetaminophen for the first 72 hours. All medications in our multimodal approach will be provided postoperatively after ACL reconstruction to both groups. The primary endpoint will be the percentage reduction in narcotics pills per patient in each group in first 72 hours postoperatively verified from sealed packages.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 15-55 years
* Primary Autograft ACL surgery
* Ability to take oral medication and willingness to patriciate in a virtual 1 and 2 week follow-up pill counts

Exclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for t the duration of the study
* Male or female, aged 15-55 years
* Primary Autograft ACL surgery
* Ability to take oral medication and willingness to patriciate in a virtual 1 and 2 week follow-up pill counts

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 30 days
  How many narcotic pills were consumed

CONTACTS AND LOCATIONS:
Overall Officials: Kurt P Spindler, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Cleveland Clinic Coral Springs, Coral Springs, Florida
  - Cleveland clinic sports medicine, Garfield, Ohio
  - Cleveland Clinic, Strongsville, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Only IPD will be used in the results publications
Supporting Information: Study Protocol, SAP
Time Frame: They will be available from the start date to the end date